CLINICAL TRIAL: NCT04456153
Title: Atovaquone for Treatment of COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Mamta K. Jain, MD,MPH, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU-2020-0707
Record Dates: First submitted 2020-06-30; First posted 2020-07-02 (Actual); Results first posted 2021-12-14 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Atovaquone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- standard of care therapy with atovaquone (Experimental): The first treatment group will receive continued standard of care therapy together with an oral dose of 1500 mg atovaquone twice daily (administered with a meal or snack) for up to 10 days.
  Interventions: Drug: Experimental Group
- standard of care therapy with matching placebo (Placebo Comparator): The second treatment group will receive continued standard of care therapy together with matching placebo.
  Interventions: Drug: Placebo Group

INTERVENTIONS:
Drug: Experimental Group — Continued standard of care therapy together with an oral dose of 1500 mg atovaquone twice daily (administered with a meal or snack) for up to 10 days
  Other Names: Atovaquone
  Arms: standard of care therapy with atovaquone
Drug: Placebo Group — Continued standard of care therapy together with matching placebo
  Arms: standard of care therapy with matching placebo

SUMMARY:
The purpose of the current study is to accelerate the use of a clinically available therapeutic already FDA-approved for other indications in the setting of pandemic COVID-19 addressing a serious and emergent unmet medical need.

This is a randomized, double-blind study of atovaquone therapy in adult participants hospitalized with COVID-19. Approximately 60 participants who meet all eligibility criteria may be randomized in a 2:1 atovaquone/placebo ratio into one of the following treatment groups:

Treatment Group 1: continued standard of care therapy together with an oral dose of 1500 mg atovaquone twice daily (administered with a meal or snack) for up to 10 days

Treatment Group 2: continued standard of care therapy together with matching placebo

DETAILED DESCRIPTION:
Design of the ATaQ COVID-19 Trial:

The purpose of the current study is to accelerate the use of a clinically available therapeutic already FDA-approved for other indications in the setting of pandemic COVID-19 addressing a serious and emergent unmet medical need. In consideration of the information included in this protocol, the overall risks to participants are outweighed by the potential benefits of atovaquone experimental therapy for the treatment of COVID-19. The benefit-risk balance for this study is considered positive.

Inclusion Criteria:

1. Diagnosis of COVID-19 by positive RT-PCR requiring hospitalization within 72 hours
2. Age ≥18 years old
3. Able to provide informed consent, or (as allowed by IRB), immediate availability of designated legally authorized representative to provide consent by proxy
4. Anticipated hospitalization for >48 hours

Exclusion Criteria

Patients who meet any of the following exclusion criteria are not to be enrolled in this study:

1. Participation in any other clinical trial with antiviral activity against COVID-19
2. Breastfeeding women
3. Known hypersensitivity to atovaquone or formulation excipient
4. Active treatment with rifampin
5. HIV patients with AIDS requiring treatment for Pneumocystis jirovecii or Toxoplasma gondii
6. Not expected to survive for 72 hours.
7. >14 days from symptom onset

   Randomization:

   Patients who meet eligibility criteria and volunteer to participate will be randomized in a 2:1 ratio to atovaquone or placebo on Day 1 using computerized randomization. An unblinded investigational pharmacist not otherwise involved in the trial will know treatment assignment and dispense investigational product. As GI absorption of atovaquone increased when taken with food, so we will administer with a meal or snack.

   Blinding:

   Double blinding of treatment assignments will be performed in this study, with the study team and patients blinded to treatment assignment.

   The list of concomitant medications will be assessed only from Day 1 prior to enrollment to Day 15 or discharge, whichever is earlier.

   Patient Enrollment and Treatment Assignment:

   Entry into screening does not guarantee enrollment into the study. In order to manage the total study enrollment, the study researchers may suspend screening and/or enrollment at any at any time.

   Pretreatment Assessments:

   Screening Visit

   Patients will be screened within 2 days before randomization and dosing to determine eligibility for participation in the study. Screening will occur under approved HIPAA waiver for research to identify and screen all hospitalized COVID-19 positive patients on a daily basis.

   Obtain informed consent.

   After informed consent has been negotiated and the form signed, the following assessments will be performed to determine eligibility requirements as specified in the inclusion and exclusion criteria:
   * Review of focused medical history including the following information (e.g., date of first symptoms, overall symptoms, exposure source, demographics, baseline characteristics), allergies and past medical history.
   * Review and record medications and therapies for the current illness
   * Recording of vital signs (heart rate, temperature, blood pressure), body weight, and height
   * Documentation of respiratory support: Respiratory Rate, Oxygen supplementation: room air, nasal canula, face mask, non-rebreather, high-flow device, mechanical ventilation; and FiO2
   * SpO2 at rest or PaO2
   * Radiographic findings

   Study patients who qualify and volunteer to participate should be immediately consented and randomized. Randomization and initiation of dosing should occur on the same day if possible.

   Baseline/Day 1 Assessments

   The following evaluations are to be completed at the Day 1 visit. The investigator must have confirmed eligibility and signing of consent before proceeding with randomization on the Day 1 visit, followed immediately by first dose of investigational product. The assessments can be completed by the patient care team and do not need to be repeated by research personnel. The following assessments must be documented before administering investigational product, using the most recent data available at the time of randomization:

   Recording of vital signs (heart rate, temperature, blood pressure, body weight, height)

   Documentation of respiratory status:

   Respiratory rate

   Oxygen supplementation and FiO2: room air, nasal canula, face mask, non-rebreather, noninvasive ventilation or high flow oxygen devices, mechanical ventilation, or ECMO

   Oxygenation: (SpO2 or PaO2)

   Radiographic findings (if available)

   Review AEs and document concomitant medications

   Document Ordinal Scale at baseline

   Obtain saliva sample and nasopharyngeal swab sample for viral load quantification at day 1 prior to initial dose

   Obtain blood for research sample

   Daily Study Assessments (Days 2-15):

   The following evaluations are to be documented daily from Days 2 - 15 or until discharge whichever comes earlier, using the data recorded at or closest to 12:00 noon each day:
   * Vital signs (heart rate, temperature, blood pressure), body weight (if available).
   * Documentation of respiratory status: Respiratory rate, Oxygen supplementation and FiO2: room air, nasal canula, face mask, non-rebreather, noninvasive ventilation or high flow oxygen devices, mechanical ventilation, or ECMO
   * Oxygenation: (SpO2 or PaO2)
   * Radiographic findings (if available)
   * Review of AEs and document concomitant medications
   * Saliva sample for COVID-19 RT-PCR every 12 hours (Days 2-8)
   * Saliva sample for COVID-19 RT-PCR once daily (Days 9-15)
   * Additional blood draws for biobanking (Day 3, and 5 only)

   Clinical Laboratory Assessments:

   Clinical laboratory assessments will be conducted as clinically indicated and all laboratory testing will be completed by local laboratories. Clinical laboratory data to be captured in the trial database will include serum chemistries, liver function tests, complete blood counts including absolute neutrophil count, hs-CRP, D-dimer, ferritin, IL-6, troponin, NTpBNP.

   SARS-CoV-2 testing will include RT-qPCR to detect or quantify SARS-CoV-2 or virus sequencing results from saliva (baseline and daily until discharge or death, and 8 days and last day of hospitalization or Day 15 if still hospitalized.

   Pretreatment and posttreatment samples with detectable SARS-CoV-2 may be sequenced for resistance monitoring of the viral polymerase gene. For all clinical laboratory tests, except those at Day 1, when more than 1 result is available in a calendar day, the value closest to 12:00 noon should be captured in the eCRF. For Day 1 tests, the most recent result before dosing should be used.

   Physical Examination:

   No physical examination is mandated by the study protocol beyond the capture of vital signs (heart rate, respiratory rate, temperature, blood pressure, SpO2 at rest or PaO2) as documented clinically.

   Post-treatment Assessments:

   Treatment will continue to complete a 10 Day course or until viral clearance is documented, whichever occurs first.

   Telephone call on Day 15 and 29 for those discharged. The phone call will include a brief survey on symptoms and information on any re-hospitalizations.

   Final review of AEs and concomitant medication.

   Vital signs will be captured if still inpatient and the ordinal scale will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of COVID-19 by positive RT-PCR requiring hospitalization within 72 hours
2. Age ≥18 years old
3. Able to provide informed consent, or (as allowed by IRB), immediate availability of designated legally authorized representative to provide consent by proxy
4. Anticipated hospitalization for >48 hours

Exclusion Criteria:

1. Participation in any other clinical trial with antiviral activity against COVID-19
2. Breastfeeding women
3. Known hypersensitivity to atovaquone or formulation excipient
4. Active treatment with rifampin
5. HIV patients with AIDS requiring treatment for Pneumocystis jirovecii or Toxoplasma gondii
6. Not expected to survive for 72 hours. 7) >14 days from symptom onset

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mamta Jain, M.D., Principal Investigator — University of Texas Southwestern Medical Center; Hesham Sadek, M.D., Principal Investigator — University of Texas Southwestern Medical Center; Ezimamaka Ajufo, M.D., Principal Investigator — University of Texas Southwestern Medical Center; Reuben Arasaratnam, M.D., Principal Investigator — University of Texas Southwestern Medical Center; James De Lemos, M.D., Principal Investigator — University of Texas Southwestern Medical Center; Helen King, M.D., Principal Investigator — University of Texas Southwestern Medical Center; Amneris Luque, M.D., Principal Investigator — University of Texas Southwestern Medical Center; Jessica Meisner, M.D., Principal Investigator — University of Texas Southwestern Medical Center; Satish Mocherla, M.D., Principal Investigator — University of Texas Southwestern Medical Center; John Schoggins, Ph.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is no specified plan made.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care Therapy With Matching Placebo | Standard of Care Therapy With Atovaquone
Started | 19 | 41
Completed | 19 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care Therapy With Atovaquone | Standard of Care Therapy With Matching Placebo | Total
Number analyzed (Participants) | 41 | 19 | 60
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 51.64 [42.5 to 60.8] | 49.4 [41 to 59.6] | 50.9 [41.9 to 59.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 7 | 22
  Male | 26 | 12 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 13 | 42
  Not Hispanic or Latino | 12 | 6 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  non-Hispanic White | 31 | 15 | 46
  Black | 6 | 2 | 8
  other | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 41 | 19 | 60
log 10 viral load (copies/mL) [Mean (Standard Deviation); unit: log 10 RNA copies/mL]
  atovaquone | 5.25 (0.278) | 0 (0) | 5.25 (0.278)
  Placebo | 0 (0) | 4.79 (0.408) | 4.79 (0.408)

OUTCOME MEASURES:

1. Primary Outcome: Primary Analysis
Description: Between group differences in viral load (Log copy number/ml) using generalized linear mixed-effect models of repeated measures (GLMM), using data from all available samples
Time Frame: Day 1 to Day 10
Population: Change in viral load from day 1 to day 10 between intervention arm and placebo
Measure: Mean (95% Confidence Interval); unit: log 10 (copies/mL)
Groups:
- Overall Group: Comparison of experimental group to placebo
- Atovaquone Group With Standard of Care Treatment: This arm received atovaquone 2: 1 in addition to the standard of care.
- Placebo Plus Standard of Care: This arm received matched placebo in addition to the standard of care.
Arm/Group | Overall Group | Atovaquone Group With Standard of Care Treatment | Placebo Plus Standard of Care
Number analyzed (Participants) | 60 | 41 | 19
log 10 (copies/mL) | -1.906 [-3.090 to 0.123] | 2.629 [1.652 to 3.606] | 4.073 [3.131 to 5.015]
Statistical Analysis 1: Comparison: Atovaquone Group With Standard of Care Treatment vs Placebo Plus Standard of Care; Test type: Superiority; p = 0.170, GLMM

2. Secondary Outcome: Secondary Between Group Differences in Viral Load
Description: Change in viral load at Day 3, 5, and 7 days. This shows the group differences between intervention and placebo and log 10 viral load at specific days 3, 5, and 7 for atovaquone arm and placebo arm.
Time Frame: baseline to day7
Measure: Mean (95% Confidence Interval); unit: log 10 (copies/mL)
Groups:
- Difference Between Atovaquone and Placebo: Comparison of experimental group to placebo
- Atovaquone Plus Standard of Care: Log 10 viral load of atovaquone group at Day 3, 5, 7
- Placebo Plus Standard of Care: Log 10 viral load of placebo group at Day 3, 5, and 7
Arm/Group | Difference Between Atovaquone and Placebo | Atovaquone Plus Standard of Care | Placebo Plus Standard of Care
Number analyzed (Participants) | 60 | 41 | 19
log 10 (copies/mL)
  day 1 to 3 | 0.129 [-0.571 to 0.829] | 5.342 [4.548 to 6.135] | 4.406 [3.609 to 5.203]
  day 1 to 5 | 0.107 [-0.610 to 0.823] | 4.329 [3.785 to 4.874] | 3.760 [2.948 to 4.572]
  day 1 to 7 | -0.766 [-1.534 to 0.002] | 3.804 [3.230 to 4.378] | 4.108 [3.270 to 4.946]
Statistical Analysis 1: Comparison: Difference Between Atovaquone and Placebo; Test type: Superiority; p = 0.051, GLMM

3. Secondary Outcome: Change in Viral Load at Day 10 Stratified by Sex
Description: Between group differences in viral load (Log copy number/ml) using GLMM stratified by
Time Frame: baseline to day 10
Population: Between group differences Day 1 to day 10
Measure: Mean (95% Confidence Interval); unit: log 10 viral load (copies/mL)
Groups:
- Stratified by Sex: Men; Stratified by Sex: Women: Comparison of change in viral load from Day 1 to day 10 between placebo and atovaquone
Arm/Group | Stratified by Sex: Men | Stratified by Sex: Women
Number analyzed (Participants) | 38 | 22
log 10 viral load (copies/mL) | -1.8732 [-3.8342 to 0.08779] | 0.555 [-1.9539 to 3.0639]

4. Secondary Outcome: Percentage With 2 Log Viral Load Drop at Day 3
Description: Between group comparison of time to drop in viral load (Log copy number/ml) of 2 log units using Kaplan-Meier estimation. Examined the percentage of participants who achieved this viral load drop in 3 days.
Time Frame: baseline to day 3
Measure: Number; unit: percentage of participants
Groups:
- Atovaquone: Atovaquone plus standard of care therapy. Proportion who had 2 log drop at Day 3
- Placebo: Matching placebo plus standard of care therapy. Proportion who had 2 log drop at Day 3
Arm/Group | Atovaquone | Placebo
Number analyzed (Participants) | 41 | 19
percentage of participants | 15 | 20

5. Secondary Outcome: Number of Participants With Change in Ordinal Scale ≥2 Points by Day 15.
Description: Ordinal scale 1 indicated death, and higher scores were various degrees of hospitalizations and incapacity to being out of hospital. Ordinal Scale 1-7 with higher score indicating improvement in clinical status. Change of ≥2 points on the ordinal scale by Day 15 using chi-square analysis
Time Frame: Day 15
Measure: Count of Participants; unit: Participants
Groups:
- Atovaquone: Atovaquone group at Day 15. Number of participants who had > or = 2 point change in ordinal score
- Placebo: Matching placebo at Day 15. Number of participants who had > or = 2 point change in ordinal score
Arm/Group | Atovaquone | Placebo
Number analyzed (Participants) | 40 | 17
Participants | 25 | 9
Statistical Analysis 1: Comparison: Atovaquone vs Placebo; Test type: Superiority; p = 0.68, Chi-squared

6. Secondary Outcome: Area Under the Curve Copies/ml*Day at Day 7
Description: This is a alternative method of measurement of area which examines the viral load ( copies/ml )(y-axis) by day (x-axis) using the trapezoidal method. The area under the curve was calculated via the trapezoidal rule. As such, this is a numeric value that is different than the traditional use of the term "mean" or "median." However, in order to calculate a measure of error associated with this quantity, bootstrapping with 500 replications would need to be performed to assess statistical significance or lack thereof. The mean of the bootstrap samples could be reported as the "mean area under the curve."
Time Frame: day 7
Measure: Number; unit: copies/mL*day
Groups:
- Atovaquone: Atovaquone plus standard of care
- Placebo: Matching placebo plus standard of care
Arm/Group | Atovaquone | Placebo
Number analyzed (Participants) | 41 | 19
copies/mL*day | 38.39 | 36.09
Statistical Analysis 1: Comparison: Atovaquone vs Placebo; Test type: Superiority; p = 0.76, trapezoidal method

7. Secondary Outcome: Stratifed by Remdesivir
Description: change in log RNA 10 day 1 to 10 stratified by remdesivir by GLMM
Time Frame: day 10
Measure: Mean (95% Confidence Interval); unit: log 10 RNA copies/mL
Groups:
- Stratified With Remdesivir: Participants who received remdesivir as part of standard of care
- Stratified Without Remdesivir: Participants who did not receive remdesivir as part of standard of care
Arm/Group | Stratified With Remdesivir | Stratified Without Remdesivir
Number analyzed (Participants) | 36 | 24
log 10 RNA copies/mL | -0.754 [-2.440 to 0.933] | -2.010 [-4.513 to 0.494]

ADVERSE EVENTS:
Time Frame: During hospitalization for an average of 10 days
Description: Collected grade 3 or 4 adverse events
Groups:
- Atovaquone: Atovaquone plus standard of care. Grade 3 and 4 adverse events were collected.
Arm/Group | Atovaquone | Placebo
All-Cause Mortality (participants affected / at risk) | 6/41 | 2/19
Serious Adverse Events (participants affected / at risk) | 7/41 | 3/19
Other Adverse Events (participants affected / at risk) | 2/41 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atovaquone (N=41) | Placebo (N=19)
hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atovaquone (N=41) | Placebo (N=19)
Transaminitis (Gastrointestinal disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was not powered for clinical endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/53/NCT04456153/Prot_SAP_000.pdf